CLINICAL TRIAL: NCT04942431
Title: REBIRTH Active School 2.0. Impact of a School-based Physical Activity Program on the Long-term Improvement of Student Health.
Brief Title: REBIRTH Active School 2.0 . a School Based Physical Activity Program
Acronym: RAS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Celine Braun, Institute for Sports Medicine, Hannover Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 7290
Record Dates: First submitted 2021-04-08; First posted 2021-06-28 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-10

CONDITIONS: Primary School Children

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventiongroup (Experimental): 60 min per day school based Physical activity program (for one year)
  Interventions: Behavioral: Rebirth active SCHOOL 2.0 movement program
- Waitinggroup (No Intervention): Intervention starts after one year.

INTERVENTIONS:
Behavioral: Rebirth active SCHOOL 2.0 movement program — 60 Minutes of physical activity per day integrated in every school-day.
  Arms: Interventiongroup

SUMMARY:
Rebirth active SCHOOL 2.0 is a physical activity intervention program and about to be realised at 40 primary schools in Lower Saxony Germany.

Half of all schools will be assigned to the intervention program or to wait for one year before starting with the movement program. After one and two years, the follow up will take place. After completing baseline examinations (i.e. physical and cognitive functions, physical activity questionnaires) the intervention program will start for one year.

The intervention program is going to be designed with the goal of implementing physical activity of 60 minutes per day. For the main module of movement impulses, the pupils will perform a 5-minute exercise in every lesson, realised by the teachers.

ELIGIBILITY:
Inclusion Criteria:

* First and second grade pupils at primary schools (District Hannover/Wolfsburg/Helmstedt/Gifhorn/Hildesheim; Lower-Saxony, Germany),

Exclusion Criteria:

* none, if no medical contraindications against intensive physical activity/tests excist.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1245 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Endurance capacity via Six-Minutes Running test | At baseline, after 1 and 2 years.
  Completed meters in Six-Minutes running test: German Motor Test 6-18 (Bös, 2009):
Change in Sprint velocity via 20 meter sprint | At baseline, after 1 and 2 years.
  20 meter sprint test measured in seconds: German Motor Test 6-18 (Bös, 2009). Scoring the best attempt out of two.
Change in Strength tests via 40 seconds of Push ups and sit ups | At baseline, after 1 and 2 years.
  Number of repetitions in 40 seconds of Push ups and sit ups: German Motor Test 6-18 (Bös, 2009)
Change in Coordination exercise: via 60 seconds Single leg stand | At baseline, after 1 and 2 years.
  Ground contacts in 60 seconds Single leg stand: German Motor Test 6-18 (Bös, 2009)

SECONDARY OUTCOMES:
Peripheral blood pressure | At baseline, after 1 and 2 years.
  Peripheral blood pressure will be measured in a seated position after a resting period of 5 minutes. We will use the oscillometric Dinamap device (Dinamap v150; Fa. GE Medical Systems, Chicago, Illinois, USA). Three measurements will be taken on the right and on the left arm. Between each measurement will be a 1 minute resting period. The Median of the left and the right arm is used for further calculations. If the Median is above the 90th percentile three measurements will be taken again by the investigator using the auscultatory method.
Central blood pressure | At baseline, after 1 and 2 years.
  Central blood pressure will be measured in a spinal position using an oscillometric device, the Mobil-O-Graph (I.E.M. GmbH). The cuff size must be chosen accordingly to the arm size. After a resting period of 5 minutes 3 measurements will be taken on the right arm. Between each measurement will be 30 seconds. The mean of the 3 measurements will be used for further calculations.
Arterial pulse wave | At baseline, after 1 and 2 years.
  Arterial pulse wave will be measured in a spinal position using the Vicorder. The patient should rest for 5 minutes before the start of the measurement. The thigh cuff will be placed around the patient's upper right thigh as high as possible. The cuff around the neck has to be placed over the right carotid artery. The investigator has to measure from the suprasternal notch vertically to the umbilicus and from the umbilicus diagonally to the mid of the thigh cuff. The length will be added up and the measurement from the suprasternal notch to the cuff around the neck will be subtracted. The length will be used for calculating the arterial pulse wave velocity. Three measurements will be taken with each having 10 consecutive waveforms with similar shape and size. The mean of the 3 measurements will be used for further calculations.
Quality of life via KidKindl | At baseline, after 1 and 2 years.
  The quality of life will be assessed applying the KidKindl questionnaire (6 questions, Likert-Skale, 24 Items, Scale 0-100) in a 1 to 1 interview. Higher scores mean a better outcome.
Physical activity questionnaire | At baseline, after 1 and 2 years.
  The physical activity will be assessed applying the physical activity questionnaire according to the KIGGS Study (MoMo Modul) in a 1 to 1 interview.
BMI (kg/m^2) | At baseline, after 1 and 2 years.
  weight and height will be combined to report BMI in kg/m^2
Body Fat Mass (kg), (%) | At baseline, after 1 and 2 years.
  Body Fat Mass will be measured in kilogram and percent via Body Impedance Measurement using the InBody 230.
Skeletal Muscle Mass (kg) | At baseline, after 1 and 2 years.
  Skeletal Muscle Mass will be measured in kilogram via Body Impedance Measurement using the InBody 230.
Fat Free Mass (kg) | At baseline, after 1 and 2 years.
  Fat Free Mass will be measured in kilogram via Body Impedance Measurement using the InBody 230.
Body height (cm) | At baseline, after 1 and 2 years.
  Measured in cm
Waist - Hip circumferences (cm) | At baseline, after 1 and 2 years.
  Measured in cm
Concentration ability | At baseline, after 1 and 2 years.
  The concentration ability will be assessed via the CCTT (children colour trail test) using the time required to perform the test and mistakes made in the test. Percentiles can be used for the comparison with peers.
Pediatric Quality of Life | At baseline, after 1 and 2 years.
  Quality of Life will be assessed via PedsQL (Quality of Life via PedsQL), 6 Questions in a 1 to 1 interview. Higher scores refect a higher quality of life.
Cognitive function | At baseline, after 1 and 2 years.
  Cognitive function (Happiness/Trust/Learning) will be assessed via questionnaire in a 1 to 1 interview (Scale 0-100, a higher score means a better outcome)
Dental health Status | At baseline, after 1 and 2 years.
  Dental health status will be assessed via questionnaire (6 Questions) in a 1 to 1 interview.
Program adherence | Whole intervention period (24 month)
  Program adherence will be assessed via Protocols by documenting the number of physical activity impulses at each participating school (minutes per day).
Phosphat (mmol/l) | At baseline, after 1 and 2 years.
  Phosphat in mmol/l will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
CysC; Cystatin C (mg/l) | At baseline, after 1 and 2 years.
  CysC in mg/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Urea (mg/dl) | At baseline, after 1 and 2 years.
  Urea in mg/dl will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Kreatinin (mg/dl) | At baseline, after 1 and 2 years.
  Kreatinin in mg/dl will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Uric acid (mg/dl) | At baseline, after 1 and 2 years.
  Uric acid in mg/dl will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
GPT; Glutamate pyruvate transaminase (U/l) | At baseline, after 1 and 2 years.
  GPT in U/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Bilirubin (mg/dl) | At baseline, after 1 and 2 years.
  Bilirubin in mg/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Triglyceride (mg/dl) | At baseline, after 1 and 2 years.
  Triglyceride in mg/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Albumin (g/l) | At baseline, after 1 and 2 years.
  Albumin in g/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
CRPhs; High-sensitivity C-reactive protein (mg/l) | At baseline, after 1 and 2 years.
  CRPhs in mg/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
HbA1c (%) | At baseline, after 1 and 2 years.
  HbA1c in % will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Cortisol (µg/l), | At baseline, after 1 and 2 years.
  Cortisol in µg/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Insulin (U/l ) | At baseline, after 1 and 2 years.
  Insulin in U/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Leukozyten (Tsd/µl) | At baseline, after 1 and 2 years.
  Leukozyten in Tsd/µl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Erythrozyten (Mio/µl) | At baseline, after 1 and 2 years.
  Erythrozyten in Mio/µl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Hb; Hemoglobin (g/dl), | At baseline, after 1 and 2 years.
  Hb in g/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Hkt;hematocrit (%) | At baseline, after 1 and 2 years.
  Hkt in %, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
MCHC ean corpuscular hemoglobin concentration (g/dl) | At baseline, after 1 and 2 years.
  MCHC in g/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Thrombozyten (Tsd/µl) | At baseline, after 1 and 2 years.
  Thrombozyten in Tsd/µl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Natrium (mmol/l) | At baseline, after 1 and 2 years.
  Natrium in mmol/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Kalium (mmol/l) | At baseline, after 1 and 2 years.
  Kalium in mmol/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Calcium (mmol/l) | At baseline, after 1 and 2 years.
  Calcium in mmol/l, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Cholesterin (mg/dl) | At baseline, after 1 and 2 years.
  Cholesterin in mg/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
HDL; High Density Lipoprotein (mg/dl) | At baseline, after 1 and 2 years.
  HDL in mg/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
LDL; Low Density Lipoprotein (mg/dl) | At baseline, after 1 and 2 years.
  LDL in mg/dl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
MCV; mean corpuscular volume (fl) | At baseline, after 1 and 2 years.
  MCV in fl, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
MCH; mean corpuscular hemoglobin (pg) | At baseline, after 1 and 2 years.
  MCH in pg, will be measured via Blood Analysis. Blood will be taken in the morning with a fasting blood test.
Urine Analysis | At baseline, after 1 and 2 years.
  Urine will be taken from the midstream urine. The children will take the sample with the help of the parents at home. The lab will measure the following urin parameters: Protein, Albumin (mg/dl), Kreatinin (g/l), Osmolarität (mOsm/kg)
Salvia Analysis | At baseline, after 1 and 2 years.
  salvia
Steps per day | At baseline, after 1 and 2 years.
  Steps per day will be assessed via Garmin Vivofit 4 devices.
Hours of sleep | At baseline, after 1 and 2 years.
  Hours of sleep will be assessed via Garmin Vivofit 4 devices.
Metabolic Equivalent | At baseline, after 1 and 2 years.
  Metabolic Equivalent (MET) (1 kcal/kg/hour) will be assessed applying Garmin Vivofit 4 devices.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Tegtbur, Prof. Dr. med., Principal Investigator — Hannover Medical School, Hannover Lower Saxony, Germany, 30625; Anette Melk, Prof. Dr. med., Principal Investigator — Medical School Hannover Lower Saxony, Germany, 30625
Locations (1):
- Hanover Medical School, Hanover, Lower Saxony, Germany